CLINICAL TRIAL: NCT02146261
Title: A Phase 1 Study of Single-dose Subcutaneous E6011 in Japanese Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E6011-J081-002
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Volunteers; Japanese; Males
MeSH Terms: interventions — quetmolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Subcutaneous administration of E6011 50 mg
  Interventions: Drug: E6011
- 2 (Experimental): Subcutaneous administration of E6011 100 mg
  Interventions: Drug: E6011
- 3 (Experimental): Subcutaneous administration of E6011 200 mg
  Interventions: Drug: E6011
- 4 (Experimental): Subcutaneous administration of E6011 400 mg
  Interventions: Drug: E6011
- 5 (Placebo Comparator): Subcutaneous administration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E6011 — Subcutaneous administration of E6011 (at doses of 50, 100, 200 and 400 mg)
  Arms: 1; 2; 3; 4
Drug: Placebo — Subcutaneous administration of placebo
  Arms: 5

SUMMARY:
This study (Protocol No. E6011-J081-002) is a single-center, randomized, double-blind, placebo-controlled, single ascending dose (SAD) study to evaluate mainly the safety and tolerability of a single subcutaneous administration of E6011. A total of 32 subjects will be randomized into four cohorts (50, 100, 200 and 400 mg groups). Of eight subjects per cohort, six subjects will receive the single subcutaneous E6011 administration and two subjects will receive the single subcutaneous placebo administration.

DETAILED DESCRIPTION:
This study consists of Screening Period, Observation Period, In-patient Period, and Follow-up Period. Screening assessments will be performed within 28 to 2 days before starting the study treatment, and Observation Period assessments will be performed on a day before starting the study treatment to confirm the eligibility of study subjects. The eligible subjects will be randomized into either E6011 arm or placebo arm using the drug allocation list prepared by the random code statistician. Each subjects dosing interval will be at least a 30-minutes.

ELIGIBILITY:
Inclusion criteria

1. Non-smoking Japanese male subjects aged greater than or equal to 20 to less than 45 years
2. BMI at screening is greater than or equal to 18.5 kg/m2 to less than 25.0 kg/m2
3. Males who have not had a successful vasectomy and their female partners must agree to practice highly effective contraception throughout the study period

Exclusion criteria

1. Has been treated with biologic product(s) (except for immunoglobulin)
2. Has received immunoglobulin or blood preparation within 6 months before the study treatment
3. Has received inoculation within 4 weeks before the study treatment
4. Has a history of autoimmune disease or immunodeficiency
5. Has a history of clinically significant angioedema, hematemesis, anal hemorrhage, or hemoptysis
6. Has a history of acute myocardial infarction, cerebral infarction, cerebral hemorrhage, or arteriosclerosis obliterans
7. With gross hematuria, occult bleeding in urine of greater than or equal to 1+ and urine protein of greater than or equal to 1+, or either of greater than or equal to 2+ is found at screening
8. Has a clinically significant vasculitis (e.g., mononeuritis multiplex)
9. Known to be positive for human immunodeficiency virus antigen/antibody (HIV antigen/antibody), hepatitis B virus surface antigen (HBs antigen), hepatitis B virus surface antibody (HBs antibody), hepatitis B core virus antibody (HBc antibody), hepatitis B virus (HBV) DNA, hepatitis C virus antibody (HCV antibody), human T cell lymphotropic virus type 1 antibody (HTVL-1 antibody), or syphilis serology test positive at screening.
10. Known to be positive for tuberculosis test (T-spot.TB Test or QuantiFERON TB Gold Test) at screening.
11. Treated with ethical drug (except for disinfectants, eye drops) within 4 weeks before the study treatment.
12. Treated with non-prescription drug (except for disinfectants, eye drops) within 2 weeks before the study treatment.
13. Has participated in another clinical trial and received an investigational drug or device within 16 weeks before the study treatment.
14. Received blood transfusion within 1 year, 400 mL or more whole blood donation within 12 weeks, or 200 mL or more whole blood donation within 4 weeks, or blood constituent donation within 2 weeks before the study treatment.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of E6011: Maximum Concentration (Cmax) | Up to 10 Weeks
Pharmacokinetics of E6011: Time to attain Cmax (tmax) | Up to 10 Weeks
Pharmacokinetics of E6011: Area Under the Concentration-time Curve From Time Zero to Time of the Last Quantifiable Concentration AUC(0-t) | Up to 10 Weeks
Pharmacokinetics of E6011: Area Under the Plasma Concentration-time Profile From Time Zero Extrapolated to Infinite Time AUC(0-inf) | Up to 10 Weeks
Pharmacokinetics of E6011: Elimination half-life (t1/2) | Up to 10 Weeks
Pharmacokinetics of E6011: CL/F | Up to 10 Weeks
  Apparent clearance of drug from plasma following extravascular administration (CL/F) was calculated as dose/AUC(0-?).
Pharmacokinetics of E6011: Apparent Volume of Distribution of Azacitidine (Vz/F) | Up to 10 Weeks
Safety and Tolerability of E6011 | Up to 10 Weeks
  The safety will be assessed based on all adverse events (AEs), clinical laboratory test, vital signs, body weight, physical finding, administration site finding, electrocardiography and chest xray.

CONTACTS AND LOCATIONS:
Locations (1):
- Sagamihara, Kanagawa, Japan